CLINICAL TRIAL: NCT00830791
Title: A Single Dose Study to Investigate the Pharmacokinetics of MK-0941 in Subjects With Renal Insufficiency
Brief Title: A Single Dose Study to Investigate the Pharmacokinetics of MK-0941 in Participants With Renal Insufficiency (MK-0941-015-02)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0941-015; 2009_522
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MK-0941 20 mg Mild Renal Insufficiency (Experimental): MK-0941 20 mg administered to participants with mild renal insufficiency and type 2 diabetes.
  Interventions: Drug: MK-0941 20 mg
- MK-0941 20 mg Moderate Renal Insufficiency (Experimental): MK-0941 20 mg administered to participants with moderate renal insufficiency and type 2 diabetes.
  Interventions: Drug: MK-0941 20 mg
- MK-0941 5 mg Severe Renal Insufficiency (Experimental): MK-0941 5 mg administered to participants with severe renal insufficiency and type 2 diabetes.
  Interventions: Drug: MK-0941 5 mg
- MK-0941 20 mg Matched Controls (Experimental): MK-0941 20 mg administered to age-, gender-, race-, body mass index (BMI)-, and hemoglobin A1C (HbAIc)-matched control subjects with normal renal function and type 2 diabetes.
  Interventions: Drug: MK-0941 20 mg
- MK-0941 5 mg Matched Controls (Experimental): MK-0941 5 mg administered to age-, gender-, race-, body mass index (BMI)-, and HbAIc-matched control subjects with normal renal function and type 2 diabetes.
  Interventions: Drug: MK-0941 5 mg

INTERVENTIONS:
Drug: MK-0941 20 mg — Two 10-mg tablets of MK-0941 administered as a single oral dose.
  Arms: MK-0941 20 mg Matched Controls; MK-0941 20 mg Mild Renal Insufficiency; MK-0941 20 mg Moderate Renal Insufficiency
Drug: MK-0941 5 mg — MK-0941 administered as one single 5-mg tablet.
  Arms: MK-0941 5 mg Matched Controls; MK-0941 5 mg Severe Renal Insufficiency

SUMMARY:
This study will assess the pharmacokinetics of MK-0941 in participants with varying degrees of renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female age 18 to 75 years
* Female of childbearing potential on appropriate method of contraception
* Body mass index (BMI) less than or equal to 40 kg/m2
* Participant is in good health
* Participant diagnosed with Type 2 Diabetes
* Participant agrees to follow smoking restrictions
* Willing to follow the study diet restrictions

Exclusion Criteria:

* Mental or legal incapacitation
* Participant has had kidney removed
* History of Type 1 diabetes
* History of stroke, chronic seizures or major neurological disorder
* History of neoplastic disease
* Nursing mother
* Consumes greater than 4 glasses of alcoholic beverages per day
* Consumes greater than 6 servings of caffeinated beverages per day
* Participant has had surgery or donated 1 unit of blood within 1 month of screening
* Participant has history of recent eye infection within 2 weeks of study drug administration
* Clinically diagnosed with glaucoma or blindness
* Has trauma to one or both eyes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941 20 mg Mild Renal Insufficiency: MK-0941 administered as a single oral dose of 20 mg (10 mg x 2) to participants with mild renal insufficiency.
- Control + MK-0941 20 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus but without mild renal insufficiency (T2DM) who received MK-941 at a dose of 20 mg administered as a single oral dose of 10 mg x 2.
- MK-0941 20 mg Moderate Renal Insufficiency: MK-0941 administered as a single oral dose of 20 mg (10 mg x 2) to participants with moderate renal insufficiency.
- Control + 20 mg MK-0941: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) but without moderate renal insufficiency who received MK-941 at a dose of 20 mg administered as a single oral dose of 10 mg x 2.
- MK-0941 5 mg Severe Renal Insufficiency: MK-0941 administered as a single oral dose of 5 mg to participants with severe renal insufficiency.
- Control + MK-0941 5 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) but without severe renal insufficiency who received MK-941 at a dose of 5 mg administered as a single oral dose.
Period: Overall Study
Arm/Group | MK-0941 20 mg Mild Renal Insufficiency | Control + MK-0941 20 mg | MK-0941 20 mg Moderate Renal Insufficiency | Control + 20 mg MK-0941 | MK-0941 5 mg Severe Renal Insufficiency | Control + MK-0941 5 mg
Started | 8 | 8 | 8 | 8 | 0 | 0
Completed | 8 | 8 | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0941 20 mg Mild Renal Insufficiency | Control + MK-0941 20 mg | MK-0941 20 mg Moderate Renal Insufficiency | Control + 20 mg MK-0941 | MK-0941 5 mg Severe Renal Insufficiency | Control + MK-0941 5 mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 0 | 32
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 |  |  | 0
  Between 18 and 65 years | 6 | 6 | 7 | 7 |  |  | 26
  >=65 years | 2 | 2 | 1 | 1 |  |  | 6
Gender [Number; unit: participants]
  Female | 6 | 6 | 5 | 5 |  |  | 22
  Male | 2 | 2 | 3 | 3 |  |  | 10

OUTCOME MEASURES:

1. Secondary Outcome: Maximum Plasma Concentration (Cmax) After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Mild Renal Insufficiency vs Matched Controls
Description: Cmax was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour CLCR of > 50 to 80 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Groups:
- MK-0941 20 mg: MK-0941 administered as a single oral dose of 20 mg (10 mg x 2).
- Control + MK-0941 20 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) who received MK-941 at a dose of 20 mg administered as a single oral dose of 10 mg x 2.
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
nM | 401.39 [230.68 to 698.43] | 543.45 [325.26 to 908.00]
Statistical Analysis 1: Comparison: MK-0941 20 mg vs Control + MK-0941 20 mg; Test type: Superiority or Other; p = 0.325, ANCOVA; Geometric Mean Ratio = 0.74, 90% CI 2-sided [0.43 to 1.26] — The mean square error on a log scale for this comparison was 0.322

2. Primary Outcome: Plasma Area Under the Curve (AUC [0-infinity]) After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Mild Renal Insufficiency vs Matched Controls
Description: Plasma AUC (0-infinity) was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency taking a single oral dose of 20 mg of MK-0941 versus controls with normal renal function taking a single oral dose of 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour creatinine clearance (CLCR) of > 50 to 80 mL/min/1.73m^2.
Time Frame: 72 Hours Post-Dose
Measure: Geometric Mean (95% Confidence Interval); unit: nM per Hour
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
nM per Hour | 1481.42 [1163.05 to 1886.93] | 1553.50 [1241.46 to 1943.98]
Statistical Analysis 1: Comparison: MK-0941 20 mg vs Control + MK-0941 20 mg; Test type: Superiority or Other; p = 0.718, ANCOVA; Geometric Mean Ratio = 0.95, 90% CI 2-sided [0.76 to 1.20] — The mean square error on a log scale was 0.061 for this comparison

3. Primary Outcome: Plasma AUC (0-infinity) After Administration of a Single Oral Dose of 20 mg of MK-0941 Among With Moderate Renal Insufficiency vs Matched Controls
Description: Plasma AUC (0-infinity) was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency taking a single oral dose of 20 mg of MK-0941 versus controls with normal renal function taking a single oral dose of 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to 50 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (95% Confidence Interval); unit: nM per Hour
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
nM per Hour | 2084.00 [1592.63 to 2726.99] | 1278.83 [987.34 to 1656.37]
Statistical Analysis 1: Comparison: MK-0941 20 mg vs Control + MK-0941 20 mg; Test type: Superiority or Other; p = 0.014, ANCOVA; Geometric Mean Ratio = 1.63, 90% CI 2-sided [1.21 to 2.20] — The mean square error on a log scale was 0.104 for this comparison

4. Primary Outcome: Plasma AUC (0-infinity) After Administration of a Single Oral Dose of 5 mg of MK-0941 Among Participants With Severe Renal Insufficiency vs Matched Controls
Description: Plasma AUC (0-infinity) was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and severe renal insufficiency taking a single oral dose of 5 mg of MK-0941 versus controls with normal renal function taking a single oral dose of 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of > 30 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Population: This study was discontinued early and participants were not treated with the 5 mg dose.
Groups:
- MK-0941 5 mg: MK-0941 administered as a single oral dose of 5 mg.
- Control + MK-0941 5 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) who received MK-941 at a dose of 5 mg administered as a single oral dose.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cmax After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Moderate Renal Insufficiency vs Matched Controls
Description: Cmax was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to 50 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
nM | 499.12 [368.13 to 676.74] | 438.57 [327.23 to 587.79]
Statistical Analysis 1: Comparison: MK-0941 20 mg vs Control + MK-0941 20 mg; Test type: Superiority or Other; p = 0.505, ANCOVA; Geometric Mean Ratio = 1.14, 90% CI 2-sided [0.81 to 1.60] — The mean square error on a log scale for this comparison was 0.133

6. Secondary Outcome: Cmax After Administration of a Single Oral Dose of 5 mg of MK-0941 Among Participants With Severe Renal Insufficiency vs Matched Controls
Description: Cmax was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and severe renal insufficiency who received 5 mg of MK-0941 versus controls with normal renal function who received 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of > 30 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Population: This study was discontinued early and participants were not treated with the 5 mg dose.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Mild Renal Insufficiency vs Matched Controls
Description: Tmax was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour CLCR of > 50 to 80 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
Hours | 1.00 [0.50 to 1.00] | 0.50 [0.50 to 2.00]
Statistical Analysis 1: Comparison: MK-0941 20 mg vs Control + MK-0941 20 mg; Test type: Superiority or Other; ANCOVA; Geometric Mean Ratio = 0.00, 90% CI 2-sided [0.00 to 0.50]

8. Secondary Outcome: Tmax After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Moderate Renal Insufficiency vs Matched Controls
Description: Tmax was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to 50 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
Hours | 0.75 [0.50 to 4.00] | 0.50 [0.50 to 2.00]
Statistical Analysis 1: Comparison: MK-0941 20 mg vs Control + MK-0941 20 mg; Test type: Superiority or Other; ANCOVA; Geometric Mean Ratio = 0.00, 90% CI 2-sided [0.00 to 0.50]

9. Secondary Outcome: Tmax After Administration of a Single Oral Dose of 5 mg of MK-0941 Among Participants With Severe Renal Insufficiency vs Matched Controls
Description: Tmax was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and severe renal insufficiency who received 5 mg of MK-0941 versus controls with normal renal function who received 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of > 30 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Population: This study was discontinued early and participants were not treated with the 5 mg dose.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time to Apparent Half Life (T 1/2) After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Mild Renal Insufficiency vs Matched Controls
Description: T 1/2 was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour CLCR of > 50 to 80 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (Standard Deviation); unit: Hours
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
Hours | 19.02 (5.45) [5.45 to 5.45] | 15.75 (7.12) [7.12 to 7.12]

11. Secondary Outcome: T 1/2 After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Moderate Renal Insufficiency vs Matched Controls
Description: T 1/2 was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency that received 20 mg of MK-0941 versus controls with normal renal function that received 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to 50 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Measure: Geometric Mean (Standard Deviation); unit: Hours
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 8 | 8
Hours | 13.59 (4.90) [4.90 to 4.90] | 11.92 (5.70) [5.70 to 5.70]

12. Secondary Outcome: T 1/2 After Administration of a Single Oral Dose of 5 mg of MK-0941 Among Participants With Severe Renal Insufficiency vs Matched Controls
Description: T 1/2 was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and severe renal insufficiency who received 5 mg of MK-0941 versus controls with normal renal function who received 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of > 30 mL/min/1.73m^2.
Time Frame: 72-Hours Post-Dose
Population: This study was discontinued early and participants were not treated with the 5 mg dose.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Amount of MK-0941 Excreted Unchanged in the Urine (Fe) After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Mild Renal Insufficiency Versus Matched Controls
Description: Fe was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour CLCR of > 50 to 80 mL/min/1.73m^2.
Time Frame: 36-Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Fe After Administration of a Single Oral Dose of 20 mg of MK-0941 Among Participants With Moderate Renal Insufficiency Versus Matched Controls
Description: Fe was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency that received 20 mg of MK-0941 versus controls with normal renal function that received 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to 50 mL/min/1.73m^2.
Time Frame: 36-Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Fe After Administration of a Single Oral Dose of 5 mg of MK-0941 Among Participants With Severe Renal Insufficiency Versus Matched Controls
Description: Fe was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency that received 5 mg of MK-0941 versus controls with normal renal function that received 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of < 30 mL/min/1.73m^2.
Time Frame: 36-Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Groups:
- Control + MK-0941 5 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) who received MK-941 at a dose of 5 mg administered as a single oral dose of 10 mg x 2.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: CLCR After Administration of a Single Oral Dose of 20 mg of MK-0941 to Participants With Mild Renal Insufficiency Versus Matched Controls
Description: CICR was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour CLCR of > 50 to 80 mL/min/1.73m^2.
Time Frame: 36-Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Groups:
- Control + MK-0941 20 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) who received MK-941 at a dose of 20 mg administered as a single oral dose (10 mg x 2).
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: CLCR After Administration of a Single Oral Dose of 20 mg of MK-0941 to Participants With Moderate Renal Insufficiency Versus Matched Controls
Description: CICR was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency that received 20 mg of MK-0941 versus controls with normal renal function that received 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to 50 mL/min/1.73m^2.
Time Frame: 36-Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: CLCR After Administration of a Single Oral Dose of 5 mg of MK-0941 to Participants With Severe Renal Insufficiency Versus Matched Controls
Description: CICR was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and severe renal insufficiency that received 5 mg of MK-0941 versus controls with normal renal function that received 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of < 30 mL/min/1.73m^2.
Time Frame: 36-Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Plasma Glucose Concentration After Administration of a Single Oral Dose of 20 mg of MK-0941 to Participants With Mild Renal Insufficiency Versus Matched Controls
Description: The glucose concentration-time profile was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and mild renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Mild renal insufficiency was defined as a 24-hour CLCR of > 50 to 80 mL/min/1.73m^2.
Time Frame: Up to 12 Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Groups:
- Control + MK-0941 20 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) who received MK-941 at a dose of 20 mg (10 mg x 2).
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Plasma Glucose Concentration After Administration of a Single Oral Dose of 20 mg of MK-0941 to Participants With Moderate Renal Insufficiency Versus Matched Controls
Description: The glucose concentration-time profile was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and moderate renal insufficiency who received 20 mg of MK-0941 versus controls with normal renal function who received 20 mg of MK-0941. Moderate renal insufficiency was defined as a 24-hour CLCR of 30 to < 50 mL/min/1.73m^2.
Time Frame: Up to 12 Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Arm/Group | MK-0941 20 mg | Control + MK-0941 20 mg
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Plasma Glucose Concentration After Administration of a Single Oral Dose of 5 mg of MK-0941 to Participants With Severe Renal Insufficiency Versus Matched Controls
Description: The glucose concentration-time profile was evaluated among participants with Type 2 Diabetes Mellitus (T2DM) and severe renal insufficiency who received 5 mg of MK-0941 versus controls with normal renal function who received 5 mg of MK-0941. Severe renal insufficiency was defined as a 24-hour CLCR of < 30 mL/min/1.73m^2.
Time Frame: Up to 12 Hours Post-Dose
Population: This study was discontinued early and this evaluation was not conducted.
Groups:
- Control + MK-0941 5 mg: Age, gender-, race-, body mass index (BMI) and hemoglobin A1C (HbA1C) matched controls with Type 2 Diabetes Mellitus (T2DM) who received MK-941 at a dose of 5 mg.
Arm/Group | MK-0941 5 mg | Control + MK-0941 5 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- MK-0941 20 mg and Mild Renal Insufficiency: MK-0941 was administered as a single oral dose to participants with mild renal insufficiency.
- MK-0941 20 mg and Moderate Renal Insufficiency: MK-0941 was administered as a single oral dose of 20 mg to participants with moderate renal insufficiency.
Arm/Group | Control + MK-0941 20 mg | MK-0941 20 mg and Mild Renal Insufficiency | MK-0941 20 mg and Moderate Renal Insufficiency
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/16 | 3/8 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control + MK-0941 20 mg (N=16) | MK-0941 20 mg and Mild Renal Insufficiency (N=8) | MK-0941 20 mg and Moderate Renal Insufficiency (N=8)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days